CLINICAL TRIAL: NCT03732235
Title: Observational Study on Transarterial Chemoembolization With Irinotecan-loaded Embolics Associated With Systemic Bevacizumab for the Treatment of Refractory Liver Metastases From Colorectal Cancer
Brief Title: TACE Associated to Systemic Bevacizumab for the Treatment of Refractory Liver Metastases From Colorectal Cancer
Acronym: EMBOBEVA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Giammaria Fiorentini (Other)
Responsible Party: Sponsor-Investigator, Giammaria Fiorentini, Dr., International Group of Endovascular Oncology
Organization: International Group of Endovascular Oncology (Other)
Other Study IDs: EMBOBEVA
Record Dates: First submitted 2018-10-30; First posted 2018-11-06 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Liver Metastasis Colon Cancer
Keywords: Liver Metastases; Transarterial chemoembolization; Bevacizumab; Anti-angiogenesis; Irinotecan; Embolics; FOLFIRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TACE+ systemic Bevacizumab: TACE was performed, using 2 ml of LifePearl® with 100 micron diameter (Terumo Europe NV, Leuven, Belgium) loaded with Irinotecan (100 mg), diluted in 5 ml of non-ionic contrast solution and 5 ml of distilled water, infused at fixed speed of 1ml/minute for a median time of 12 minutes (range 8-16 minutes). A second TACE was performed after 30 days if needed according to physician choice.
  Bevacizumab (5 mg/kg) therapy was initiated 15 days after first round of TACE and was repeated every two weeks, for a total of 8 cycles.
  Interventions: Device: TACE+ systemic Bevacizumab
- FOLFIRI+Bevacizumab: FOLFIRI consists of 5-FU administered as a 48-hour continuous infusion to a total dose of 3,200 mg/m2 without a bolus, leucovorin 200 mg/m2, irinotecan 165 mg/m2 Bevacizumab (5 mg/kg) therapy was repeated every two weeks, for a total of 8 cycles.
  Interventions: Drug: FOLFIRI+Bevacizumab
- TACE: TACE was performed, using 2 ml of LifePearl® with 100 micron diameter (Terumo Europe NV, Leuven, Belgium) loaded with Irinotecan (100 mg), diluted in 5 ml of non-ionic contrast solution and 5 ml of distilled water, infused at fixed speed of 1ml/minute for a median time of 12 minutes (range 8-16 minutes). A second TACE was performed after 30 days if needed according to physician choice.
  Interventions: Device: TACE

INTERVENTIONS:
Device: TACE+ systemic Bevacizumab — PEG embolics
  Groups: TACE+ systemic Bevacizumab
Drug: FOLFIRI+Bevacizumab — antiangiogenic factor
  Groups: FOLFIRI+Bevacizumab
Device: TACE — PEG embolics
  Groups: TACE

SUMMARY:
Transarterial chemoembolization (TACE) is an effective, minimally invasive therapy that is widely used for unresectable colorectal cancer liver metastases (CRC-LM) treatment. Chemoembolization, however, induces a hypoxic micro-environment, which increases neo-angiogenesis, and may promote early progression. For this reason, efficacy may be improved by associating TACE with an angiogenesis inhibitor, such as bevacizumab.

The use of FOLFIRI associate to Bevacizumab is part of clinical practice and is commonly used for the therapy of patients with CRC-LM both wild type and mutant.

This case-control observational study aim to compare patients treated with TACE using Irinotecan-loaded embolics followed by systemic Bevacizumab versus patients treated with FILFIRI+ Bevacizumab

DETAILED DESCRIPTION:
TACE is indicated for the treatment of unresectable CRC_LM, patients who are refractory to systemic chemotherapy, elderly, or have a poor performance status, and is usually performed using irinotecan (IRI) covalently loaded onto embolics.

Although chemoembolization with irinotecan-loaded embolics results in an objective response, this method creates a hypoxic micro-environment. Hypoxia induces and activates the HIF-1 and HIF 2 hypoxia-inducible transcription factors, which promote high-level VEGF expression and subsequent neo-angiogenesis.

This may provide a mechanism for early relapse and progression following TACE and strongly support a rational for following TACE therapy with a therapeutic inhibitor of angiogenesis, such as bevacizumab.

The use of FOLFIRI associate to Bevacizumab is part of clinical practice and is commonly used for the therapy of patients with CRC-LM both wild type and mutant.

This case-control observational study aim to compare patients treated with TACE using Irinotecan-loaded embolics followed by systemic Bevacizumab versus patients treated with FILFIRI+ Bevacizumab

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* >18 years old;
* diagnosed with unresectable CRC-LM (for reasons of anatomy, co-morbidity, patient's wishes, lack of response to standard therapy with intravenous or oral fluoropyrimidine, oxaliplatin, irinotecan or biological agents (bevacizumab, cetuximab, panitumumab);
* Eastern Cooperative Oncology Group (ECOG) 0-1;
* measurable tumor size by mRECIST [6];
* ≤40% liver involvement;
* a life expectancy of at least 3 months,
* blood biochemistry within the normal range.

Exclusion Criteria:

* contraindication for angiographic catheterization;
* extensive extra-hepatic disease;
* pregnancy or breast-feeding,
* other severe clinical contraindications (e.g. liver failure, ascites, cardiovascular diseases and/or chronic obstructive pulmonary disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a prospective observational single center study.that involved CRC-LM patients treated with TACE, using irinotecan-loaded PEG embolics (LIFIRI), followed by the intravenous administration of bevacizumab. This group was compared to CRC-LM patients treated with FOLFIRI+Bevacizumab.
  CRC-LM patients were instructed by physician about the study procedures and after signing informed consent choose the type of theratment TACE+bevacizumab or FOLOFIRI+bevacizumab
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
time to progression | 1 year
  time from first treatment to progression will be computed

SECONDARY OUTCOMES:
Tumor response | 3 months
  CT scan will be performed to assess tomuor response
Number of adverse events | 3 motnhs
  Number of adverse events will be monitored

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Ospedali Riuniti Marche Nord, Presidio Ospedaliero San Salvatore, Pesaro, PU, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be shared
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: request by email to Principal Investigator

REFERENCES:
- [Derived] Fiorentini G, Sarti D, Nardella M, Inchingolo R, Nestola M, Rebonato A, Guadagni S. Chemoembolization Alone or Associated With Bevacizumab for Therapy of Colorectal Cancer Metastases: Preliminary Results of a Randomized Study. In Vivo. 2020 Mar-Apr;34(2):683-686. doi: 10.21873/invivo.11824. PMID 32111770